CLINICAL TRIAL: NCT06258421
Title: Burden of Disease and Living Situation in Desmoid Patients
Acronym: PROSa Desmoid
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: SOS Desmoid e.V. (Unknown); Universitätsmedizin Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: SR+BO-EK-388092023
Record Dates: First submitted 2024-01-24; First posted 2024-02-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-02

CONDITIONS: Desmoid Tumor; Quality of Life
Keywords: Health-related Quality of Life; Unmet needs; Return to normal life
MeSH Terms: conditions — Desmoid Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Desmoid Tumor Patients: People who have been diagnosed with a desmoid tumor after the age of 18
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Observatory Study

SUMMARY:
The main aim of the study is to assess the situation and quality of life of desmoid patients. Impaired areas of quality of life and the associated factors are to be identified. The survey is planned as a cross-sectional study (patient survey).

Prevalent and incident desmoid patients will be identified at the University Hospital Mannheim and checked for eligibility. Quality of life and patient-reported data are collected by means of written questionnaires. Medical data is collected from patient files in the clinics. The aim is to include 100 patients. Descriptive analyses of the variables collected and regression models are planned as statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Desmoid diagnosis (primary neoplasia, all stages)
* Age ≥18 years at diagnosis

Exclusion Criteria:

* Inability to complete a structured questionnaire (insufficient language skills; dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have been diagnosed with a desmoid tumorafter the age of 18. Treatment at the Mannheim University Hospital or via SOS Desmoid e.V.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life (EORTC C30) | baseline
  Health-Related Quality of Life Questionnaire

SECONDARY OUTCOMES:
The Brief Pain Inventory (BPI) | baseline
  The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Reintegration to Normal Living (RNL) Index | baseline
  Reintegration to normal living as a proxy to quality of life
Supportive Care Needs Survey | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martin Eichler, Dr., M.Sc. / PHD, Principal Investigator — Universitätsklinikum Carl-Gustav-Carus Dresden
Locations (1):
- Universitätsklinikum Carl-Gustav-Carus Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No